CLINICAL TRIAL: NCT05995002
Title: Effects of Increasing Anthocyanin Intake on Cardiometabolic Biomarkers in Patients With Coronary Artery Disease
Brief Title: Anthocyanin Intake on Cardiometabolic Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Nasrollahzadeh, Associate Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 43004233
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Stenosis
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Conventional drug treatment with a general recommendation for a healthy diet.
- Anthocyanin-rich diet group (Experimental): Conventional drug treatment with a weekly food plan aims to increase the consumption of anthocyanin-rich sources
  Interventions: Other: Anthocyanin-rich diet

INTERVENTIONS:
Other: Anthocyanin-rich diet — A weekly food plan aims to increase the consumption of anthocyanin-rich sources such as berries, black grapes (or currants), cherries, strawberries, pomegranates, and red onions.
  Arms: Anthocyanin-rich diet group

SUMMARY:
Flavonoids are one of the main groups of polyphenols. Anthocyanins, which are a subgroup of the flavonoid family, are found in a number of fruits and some vegetables. In epidemiological studies, high dietary intake of polyphenols has been associated with improvement of some cardiometabolic risk factors in high-risk individuals. Furthermore, in controlled studies, consumption of polyphenol-rich food sources or anthocyanin extract supplementation has improved some cardiometabolic factors. In the present study, the effect of diet enriched with anthocyanin-rich food sources on cardiometabolic factors will be studied in coronary artery disease patients.

DETAILED DESCRIPTION:
This study is an unblinded randomized controlled clinical trial. In this study, among the patients referred to Shahid Modares Hospital (Tehran, IRAN), those who are willing to participate and have inclusion criteria will be recruited. Inclusion criteria are coronary heart disease with recent coronary angiography, age range of 30-75 years. Exclusion criteria are end-stage renal disease, patients undergoing chemotherapy or radiotherapy, patients with inflammatory bowel syndrome, patients being treated with glucocorticoid drugs or antibiotics. Patients are randomly assigned to one of two study groups, including the control group and the group consuming food sources rich in anthocyanin in the diet. The duration of the study will be 8 weeks. In the control group, a general recommendation related to a healthy diet such as reducing the intake of saturated fats, sodium, and simple sugars, is provided. In the anthocyanin-rich diet group, the weekly food plan aims to increase the consumption of anthocyanin-rich sources such as berries, black grapes (or currants), cherries, strawberries, pomegranates, and red onions. The patients' drug regimen will not change during the study. Patients are asked not to use over-the-counter herbal medicines and nutritional supplements during the study. At the beginning and end of the study, blood,

ELIGIBILITY:
Inclusion Criteria:

* coronary heart disease with recent coronary angiography

Exclusion Criteria:

* End-stage renal disease,
* Patients undergoing chemotherapy or radiotherapy,
* Patients with inflammatory bowel syndrome
* Patients being treated with glucocorticoid drugs or antibiotics.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Plasma inflammatory factors concentration | 8 weeks
  fasting plasma concentration of C-reactive protein and IL-6

SECONDARY OUTCOMES:
Plasma concentration of insulin | 8 weeks
  Fasting plasma concentration of insulin
Plasma levels of lipids and lipoproteins | 8 weeks
  Fasting plasma levels of triglycerides, HDL-cholesterol, and LDL-cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- Shahid Modares Hospital, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: No